CLINICAL TRIAL: NCT02900300
Title: Constitution of a Biobank to Optimize in Vitro an Antioxydant Treatment for Diaphragm Dysfunction Induced by Mechanical Ventilation
Brief Title: A Biobank for Diaphragm Muscular Fiber
Acronym: BOTAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL15_0389
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Diaphragm Dysfunction; Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Diaphragmatic muscle collected during a digestive surgery for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm from the care will be conserved.
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study focuses on mechanical ventilation used in intensive care unit to supplement ventilatory function in patients. Mechanical ventilation can "paradoxically" be at the origin of complications that can be life-threatening in patients. This muscular pathology is called ventilation-induced diaphragmatic dysfunction (DDIV).

Diaphragmatic muscle collected during a digestive surgery for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm from the care will be conserved. The diaphragm biopsy from the care will be retained for biobanking to obtain myoblast in culture which will differentiate in Diaphragm fiber. Then these fibers will be submitted under mechanical stress condition similar to those imposed in vivo by mechanical ventilation to validate in human a model in vitro of diaphragm dysfunction induced by mechanical ventilation. Then the second part of the study will be to evaluate with this model, the efficiency of an antioxidant therapy.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 65 years old
* patient treated by the digestive surgery department of Montpellier University Hospital for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm
* Non-smoker patient for more than 6 months
* patient clinically stable at the time of the study, ie not requiring any treatment

Exclusion Criteria:

* Patients undergoing treatment with antibiotics or corticosteroids, or recently within the last 4 months
* Patients with a body mass index > 30
* Patients with any criteria that may in themselves impair respiratory muscle function such as chronic obstructive pulmonary disease, heart failure, systemic infection, neuromuscular pathology, psychiatric pathology or metabolic disorder.

Patients with coagulopathy or thrombocytopenia.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing a surgery for a benign or malignant tumor of the liver requiring surgical excision in contact with the diaphragm
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Myoblast differentiation capacity | 24 month
  Description: evaluation of ROS (reactive oxygen species) production by confocal microscopie of diaphragm fiber submitted in vitro by mechanical stress.

SECONDARY OUTCOMES:
Myoblast proliferation capacity | 24 month
  Description: Evaluation of diaphragm myoblast differenciation capacity in vitro under different concentration of antioxydant.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided